CLINICAL TRIAL: NCT02769390
Title: Association of Different Doses of Clonidine in Caudal Epidural Anesthesia for Hypospadias Surgery
Acronym: clonidine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAAE23332313600005149
Record Dates: First submitted 2015-04-09; First posted 2016-05-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Pain
Keywords: Analgesia; Bupivacaine; Clonidine
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Clonidine; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bupivacaine 0,166% (No Intervention): General Anesthesia associated with caudal anesthesia with Bupivacaine 0,166% for hypospadia surgery
- Clonidine 1 mcg/Kg (Active Comparator): IGeneral Anesthesia associated with caudal anesthesia with Bupivacaine 0,166% plus 1 mcg/ Kg of clonidine for hypospadia surgery
  Interventions: Drug: Clonidine 1 mcg/Kg
- Clonidine 2 mcg/ Kg (Active Comparator): IGeneral Anesthesia associated with caudal anesthesia with Bupivacaine 0,166% plus 2 mcg/ Kg of clonidine for hypospadia surgery
  Interventions: Drug: Clonidine 2 mcg/ Kg
- Clonidine 3 mcg/Kg (Active Comparator): General Anesthesia associated with caudal anesthesia with Bupivacaine 0,166% plus 3 mcg/ Kg of clonidine for hypospadia surgery
  Interventions: Drug: Clonidine 3 mcg/ Kg

INTERVENTIONS:
Drug: Clonidine 1 mcg/Kg — Clonidine 1 mcg/Kg associated with bupivacaine 0,166% 1 ml/Kg administred epidural caudal in children for hypospadias surgery
  Other Names: Atensine
  Arms: Clonidine 1 mcg/Kg
Drug: Clonidine 2 mcg/ Kg — Clonidine 2 mcg//Kg associated with bupivacaine 0,166% 1 ml/Kg administred epidural caudal in children for hypospadias surgery
  Other Names: Atensine
  Arms: Clonidine 2 mcg/ Kg
Drug: Clonidine 3 mcg/ Kg — Clonidine 3 mcg //Kg associated with bupivacaine 0,166% 1 ml/Kg administred epidural caudal in children for hypospadias surgery
  Other Names: Atensine
  Arms: Clonidine 3 mcg/Kg

SUMMARY:
The use of increasing doses of clonidine ssociated to bupivacaine in caudal epidural block provides better postoperative analgesia compared whit analgesia provide by bupivacaine alone

It is a randomized, double blind study, involving 80 children with ages from 1 to 10 years old, following eletive hypospadias surgery, under general anesthesia and caudal epidural block . The patients will be divided into 4 groups: bupivacaine alone, bupivacaine plus clonidine 1mcg/kg, bupivacaine plus clonidine 2 mcg/kg, bupivacaine plus clonidine 3 mg/kg. The peroperative consumption of anesthetics gases, heart rate and arterial blood pressure will be recorded. Postoperative pain will be evaluated by using FLACC scale ( faces , legs, activity , cry , consolability ) . Requiriments for supplementary postoperative analgesia at 24 h will be avaiable.

DETAILED DESCRIPTION:
It is a randomized, double blind study, involving 80 children with ages from 1 to 10 years old, following eletive hypospadias surgery, under general anesthesia and caudal epidural block . The patients will be divided into 4 groups: bupivacaine alone, bupivacaine plus clonidine 1mcg/kg, bupivacaine plus clonidine 2 mcg/kg, bupivacaine plus clonidine 3 mg/kg. The peroperative consumption of anesthetics gases, heart rate and arterial blood pressure will be recorded. Postoperative pain will be evaluated by using FLACC scale ( faces , legs, activity, cry , consolability ) . Requiriments for supplementary postoperative analgesia at 24 h will be avaiable. Postoperative hemodynamics parameters will be recordes at 24 h.

ELIGIBILITY:
Inclusion Criteria:

* CHildren 1 - 10 years old.
* ASA I E II ( American Society of Anesthesiology)
* hypospadias surgery

Exclusion Criteria:

* parents refuse
* Infection
* Coagulation disorders
* Allergy to anesthetics
* Abnormalities of the sacral spine

Ages: 1 Year to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Analgesia and efficacy of a bupivacaine-clonidine mixture measured through postoperative morphine consumption | 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: ana claudia mota bonisson, M, Principal Investigator — Hospital da Baleia - Fundação Benjamim Guimaraes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes ML, Pires KC, Tiburcio MA, Gomez RS. Caudal bupivacaine supplemented with morphine or clonidine, or supplemented with morphine plus clonidine in children undergoing infra-umbilical urological and genital procedures: a prospective, randomized and double-blind study. J Anesth. 2012 Apr;26(2):213-8. doi: 10.1007/s00540-011-1297-y. Epub 2011 Dec 10. PMID 22159880
- [Background] Mauch J, Weiss M. [Pediatric caudal anesthesia: importance and aspects of safety concerns]. Schmerz. 2012 Aug;26(4):443-53; quiz 454. doi: 10.1007/s00482-012-1202-0. German. PMID 22855315